CLINICAL TRIAL: NCT05387720
Title: Concurrent Trigger Sensitivity Adjustment And Diaphragmatic Facilitation On Weaning Of Patients From Mechanical Ventilation
Brief Title: Concurrent Trigger Sensitivity Adjustment And Diaphragmatic Facilitation On Weaning From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Badran Mohamed Ismail, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002902
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Acute Respiratory Failure; Mechanically Ventilated Patients
Keywords: Acute Respiratory Failure; Mechanical ventilation; Ventilator Induced diaphragmatic dysfunction; Proprioceptive neuromuscular training; Diaphragmatic facilitation; Diaphragmatic PNF; Inspiratory Muscle training; Trigger sensitivity
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group A (Active Comparator): Study Group A (25 patients) will receive manual diaphragmatic facilitation (PNF) technique in addition to traditional chest physiotherapy
  Interventions: Procedure: Manual diaphragmatic facilitation (PNF) technique
- Study Group B (Active Comparator): Study Group B (25 patients) will receive trigger sensitivity adjustment on mechanical ventilator in addition to traditional chest physiotherapy.
  Interventions: Procedure: Trigger sensitivity adjustment on mechanical ventilation
- Study Group C (Active Comparator): Study Group C (25 patients) will receive a concurrent trigger sensitivity adjustment and manual diaphragmatic facilitation (PNF) technique in addition to traditional chest physiotherapy.
  Interventions: Procedure: concurrent trigger sensitivity adjustment and manual diaphragmatic facilitation (PNF) technique

INTERVENTIONS:
Procedure: Manual diaphragmatic facilitation (PNF) technique — Diaphragmatic PNF is a facilitator technique used to improve chest expansion, increase epigastric excursion, promote breathing frequency and depth, by applying external proprioceptive tactile stimuli over diaphragm. The therapist places the thumbs toward the xiphoid process and the fingers along the costal margins of the lower ribs and pushing deep to stimulate the diaphragm During inspiration, the patient will be instructed "take a deep breath breathe in" and the therapist assists the movement to promote the subject's respiratory pattern in downward movement. At the maximum inspiration, therapist will say "hold your breath for 5 seconds". The therapist gives mild resistance to the inferior movement of the contracting diaphragm during inspiration while pushing diaphragm superiorly. During expiration, therapist says "breathe out" and pushed under lower ribs on both sides upward to assist the discharge of air remaining in the lungs.
  Other Names: Diaphragmatic PNF
  Arms: Study Group A
Procedure: Trigger sensitivity adjustment on mechanical ventilation — The pressure trigger sensitivity will be adjusted to 20% of the first recorded MIP at the start of training by decreasing trigger sensitivity towards negative pressure. In the first session, inspiratory muscle training (IMT) will be limited to 5 min; afterwards the duration will be increased by 5 min at every session until it reaches 30 min. If a patient tolerates 30 min of IMT, The next session will be performed with increasing negative pressure of the trigger sensitivity by 10% of the initial MIP. The maximal acceptable intensity is 40% of MIP, Patients who can't tolerate IMT with 20% of MIP for 5 min will be trained with 10% of MIP
  Other Names: Trigger sensitivity
  Arms: Study Group B
Procedure: concurrent trigger sensitivity adjustment and manual diaphragmatic facilitation (PNF) technique — Diaphragmatic PNF technique will be applied synchronously in the same time, on each breath with trigger sensitivity adjustment on mechanical ventilation in same manner as discussed before
  Arms: Study Group C

SUMMARY:
As Acute respiratory failure (ARF) is a challenging serious condition especially when it necessitates intubation to deliver mechanical ventilation which is a fundamental strategy for supporting the respiratory function when the patient can't bear all work of breathing. Even if it represents a life-saving procedure, mechanical ventilation (MV) is associated to life-threatening complications as respiratory muscle dysfunction, and atrophy that lead to long stay in intensive care unit (ICU) and higher mortality. Weaning difficulty is experienced in nearly 30 percent of critically ill patients.

The decision to extubate mechanically ventilated patients should be aimed at preventing both the risk of premature liberation from MV which is associated with poor outcome and the risk of delayed extubation which increases the complications of prolonged MV and there is increasing evidence that MV itself may adversely affect the diaphragm's structure and function, which has been termed ventilator-induced diaphragmatic dysfunction (VIDD). The combination of positive pressure ventilation and positive end-expiratory pressure may unload the diaphragm which leads to changes in myofibril length and rapid atrophy that occurs within hours of MV, caused by an imbalance between protein synthesis and proteolysis, lead to a large reduction in the inspiratory pressure generated by the diaphragm.

DETAILED DESCRIPTION:
Physiotherapist is a key member of multidisciplinary team and plays an vital role in ICU in improving the patient's quality of life, Inspiratory muscle training (IMT) applies a load to the diaphragm and accessory inspiratory muscles to increase their strength and endurance. Adjustment of ventilator sensitivity provides resistance and hence a pressure load to the inspiratory muscles, and proprioceptive neuromuscular facilitation (PNF) of respiration is newly introduced in ICU for patients who are ventilator dependent by use of external proprioceptive and tactile stimuli to assist respiration. PNF techniques improve inspiration and expiration in next cycle that shows improvement with active initiation or more participation in respiration to alter the rate and depth of breathing, facilitate respiratory muscles, improve breathing pattern and increase tidal volume So the purpose of this study is to determine the concurrent effect of trigger sensitivity adjustment and diaphragmatic facilitation on weaning of patients from mechanical ventilation. As the patients may gain a more benefit from the combination of trigger sensitivity adjustment and manual diaphragmatic facilitation (PNF) techniques than from each one alone. Therefore, a concurrent trigger sensitivity adjustment and manual diaphragmatic facilitation (PNF) techniques must likely be started within 24 to 48 hours of initiating MV to protect diaphragm from atrophy, facilitate faster weaning, minimize ICU stay and cost of treatment, and decrease the morbidity and mortality rate of those patients admitted to ICU.

Study Hypothesis:

It will be hypothesized that there is no effect of diaphragmatic facilitation on weaning of patients from mechanical ventilation.

It will be hypothesized that there is no effect of trigger sensitivity adjustment on weaning of patients from mechanical ventilation.

It will be hypothesized that there is no effect of a concurrent trigger sensitivity adjustment and diaphragmatic facilitation on weaning of patients from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with age ranges (50-60) years old.
* Patients will be referred with acute respiratory failure (ARF) inside ICU.
* All patients are intubated and mechanically ventilated with assisted control (pressure or volume) or pressure support modes for 24-48 hours.
* All patients with positive end expiratory pressure (PEEP) don't exceed 10 cmH2o.
* All patients are hemodynamically stable; temperature (36.2-37.5) C, Heart rate < 140 /min, Blood pressure (systolic: <180mmHg and diastolic <100 mmHg), Respiratory rate < 35/min and oxygen saturation >90%
* All patients are conscious and responsive to verbal command.

Exclusion Criteria:

* Fraction of inspired oxygen (fio2)>0.6 and SPO2 < 85% to avoid further hypoxia and respiratory distress.
* Positive end expiratory pressure (PEEP) > 10 cmH2O to avoid barotrauma.
* Severe pulmonary condition; acute pulmonary embolism, undrained pneumothorax.
* Unstable hemodynamic condition as defined by heart rate more than 140 beats/min, systolic blood pressure >180 mmHg or Low blood pressure < 80 mmHg and respiratory rate is exceeding 35 breaths/min.
* Patients who develop any cardiac condition during the course of treatment; acute myocardial infarction or cardiac arrhythmia.
* Patients who recently have undergo cardiac or abdominal or gynecological surgery.
* Active lung infection like tuberculosis.
* Chest trauma such as rib fracture, flail chest, thoracic vertebra fracture or chest burns.
* Spinal cord injuries involved the phrenic nerve.
* Active bleeding as alveolar hemorrhage, hemoptysis.
* Heavy sedation that depresses respiratory drive or ability to follow commands.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Blood gases analysis | Blood gases will be analyzed and recorded for all patients pre and post the treatment program duration 5 up to 7 days
  Blood gases analyzer(SIEMENS RAPIDLAB 1265, manufactured in 2008) is used in every clinical diagnosis lab or critical care facility to measure blood gases (PH, pco2 and po2), electrolytes, and metabolites parameters from whole blood samples. An arterial blood catheter (cannula) was inserted into the radial artery to draw blood sample of (2 to 3) ml, in a (3 to 5) ml plastic airtight syringe fitted with a small bore needled and filled with heparin.
  The standard values: PH 7.35-7.45, PaCO2 35-45, PaO2 60-100, SPO2 95-100% and PaO2/FiO2 ratio >300.
Oxygenation Index (OI) | OI will be recorded for three study groups pre and post the treatment program duration 5 up to 7 days
  OI is recognized as the primary indicator for respiratory disease severity stratification in mechanically ventilated patients to assess the intensity of ventilatory support that needed to maintain adequate oxygenation and predict outcomes in patients with ARF.
  OI = (FiO2 x MAP) / PaO2 OI normally, <15 as the lower the OI the better the outcome: as the oxygenation of the patient improves, they can achieve a higher PaO2 at a lower FiO2.
Maximum Inspiratory Pressure (MIP) | MIP will be measured digitally from the MV for all patients pre and post the treatment program duration 5 up to 7 days.
  MIP also known as negative inspiratory force (NIF); the maximum negative pressure generated for at least 1 second during maximal inspiratory effort against occluded airway that estimated inspiratory muscle strength mainly diaphragm. PImax has been widely used to quantify respiratory muscle weakness. PImax values of more than -25 cmH2O was considered as an index to predict weaning success.
  To obtain reliable results, the maneuver will be performed three times, with a 1-min interval between readings. The highest value was chosen as PImax.
Rapid shallow breathing index (RSBI) | RSBI was measured for all patients pre and post the treatment program duration 5 up to 7 days
  RSBI is an index used to predict weaning from MV, defined as the ratio of respiratory frequency to tidal volume (f/VT). People on MV who cannot tolerate independent breathing tend to breath rapidly (high frequency) and shallowly (low tidal volume) and will therefore have a high RSBI. RSBI<105 is reported to be the most accurate predictor of successful patient extubation.
  ventilator mode was switched on CPAP with zero pressure support to divide f by Vt to obtain RSBI (f/Vt).
Weaning Success Rate | it will be recorded for three study groups post the treatment program duration 5 up to 7 days
  Weaning success is defined as spontaneous breathing without mechanical support for at least 48 hours. Weaning success rate (a proportion of successfully weaned patients to total number of patients receiving a treatment program)

CONTACTS AND LOCATIONS:
Overall Officials: Hany E Obaya, PHD, Study Chair — Cairo University; El sayed E El sayed, PHD, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy - Cairo University, Giza, Egypt